CLINICAL TRIAL: NCT01057251
Title: Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Effect of 5 mg or 20 mg Nebivolol Once Daily on Blood Pressure in Patients With Systolic Stage 2 Hypertension
Brief Title: Nebivolol in Patients With Systolic Stage 2 Hypertension
Acronym: NEB-MD-20
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEB-MD-20
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Results first posted 2012-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2011-12

CONDITIONS: Hypertension
Keywords: Nebivolol; Bystolic TM; Hypertension; Stage 2 Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nebivolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Nebivolol
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nebivolol — 5 mg, titrated to 20 mg, once daily oral administration
  Other Names: Bystolic
  Arms: 1
Drug: Placebo — 5 mg or 20 mg once daily, oral administration
  Arms: 2

SUMMARY:
The primary object of this study is to evaluate the efficacy and safety of 6 weeks of nebivolol monotherapy compared with placebo in patients with systolic stage 2 hypertension.

ELIGIBILITY:
Inclusion Criteria:

* male of female, 18 to 64 years of age at screening
* mean seated heart rate at least 60 bpm
* diagnosed systolic stage 2 hypertension
* unremarkable physical exam findings

Exclusion Criteria:

* high risk due to secondary hypertension or former stage 3 hypertension by JNC6
* concurrent conditions (reno, cardiovascular, obesity, thyroid, etc)
* currently taking medication that cannot be stopped during the course of the study
* participating other clinical trials
* member of the study center personnel
* documented drug abuse
* contra indication to beta blocker
* abnormal lab finding
* poor compliance
* other conditions judged by investigator that is not suitable for the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 433 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Stapff, MD, PhD, Study Director — Forest Research Institute, a Subsidiary of Forest Laboratories Inc.
Locations (36):
- United States (36):
  - Forest Investigative Site 008, Foley, Alabama
  - Forest Investigative Site 021, Montgomery, Alabama
  - Forest Investigative Site 006, Chino, California
  - Forest Investigative Site 002, Long Beach, California
  - Forest Investigative Site 004, Los Angeles, California
  - Forest Investigative Site 020, Temecula, California
  - Forest Investigative Site 028, Coral Gables, Florida
  - Forest Investigative Site 014, Daytona Beach, Florida
  - Forest Investigative Site 001, Fort Lauderdale, Florida
  - Forest Investigative Site 037, Fort Lauderdale, Florida
  - Forest Investigative Site 033, Hialeah, Florida
  - Forest Investigative Site 026, Jacksonville, Florida
  - Forest Investigative Site 017, Miami, Florida
  - Forest Investigative Site 010, Miami, Florida
  - Forest Investigative Site 030, Orlando, Florida
  - Forest Investigative Site 009, Atlanta, Georgia
  - Forest Investigative Site 031, Augusta, Georgia
  - Forest Investigative Site 039, Meridian, Idaho
  - Forest Investigative Site 007, Auburn, Maine
  - Forest Investigative Site 038, Baltimore, Maryland
  - Forest Investigative Site 011, Baltimore, Maryland
  - Forest Investigative Site 029, Prince Frederick, Maryland
  - Forest Investigative Site 023, Paw Paw, Michigan
  - Forest Investigative Site 005, Florissant, Missouri
  - Forest Investigative Site 041, Las Vegas, Nevada
  - Forest Investigative Site 040, New York, New York
  - Forest Investigative Site 012, Hickory, North Carolina
  - Forest Investigative Site 027, Salisbury, North Carolina
  - Forest Investigative Site 024, Harleysville, Pennsylvania
  - Forest Investigative Site 013, Charleston, South Carolina
  - Forest Investigative Site 035, Greenville, South Carolina
  - Forest Investigative Site 018, Mt. Pleasant, South Carolina
  - Forest Investigative Site 022, Simpsonville, South Carolina
  - Forest Investigative Site 003, Memphis, Tennessee
  - Forest Investigative Site 032, Corpus Christi, Texas
  - Forest Investigative Site 025, Richmond, Virginia

REFERENCES:
- [Derived] Lewin A, Punzi H, Luo X, Stapff M. Nebivolol monotherapy for patients with systolic stage II hypertension: results of a randomized, placebo-controlled trial. Clin Ther. 2013 Feb;35(2):142-52. doi: 10.1016/j.clinthera.2012.12.015. Epub 2013 Jan 15. PMID 23332366

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occured from March 2010 through October 2010 at 36 US sites.
Pre-assignment Details: A 4 week single-blind placebo washout phase was required for patients on anti-hypertensives at screening.
Groups:
- Placebo: Dose-matched placebo, once daily oral administration
Period: Overall Study
Arm/Group | Nebivolol | Placebo
Started | 290 | 143 (The safety population is 142, as one patient was randomized, but never received study drug.)
Completed | 262 | 114
Not Completed | 28 | 29
Not completed — Did not meet InclusionExclusion criteria | 4 | 2
Not completed — Adverse Event | 4 | 2
Not completed — Lack of Efficacy | 2 | 11
Not completed — Protocol Violation | 6 | 2
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 7 | 6
Not completed — Other Reason | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Placebo | Total
Number analyzed (Participants) | 290 | 142 | 432
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 290 | 142 | 432
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 51.1 (8.1) | 49.7 (9.0) | 50.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 61 | 202
  Male | 149 | 81 | 230
Region of Enrollment [Number; unit: participants]
  United States | 290 | 142 | 432

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Seated Systolic Blood Pressure After 6 Weeks of Nebivolol Monotherapy
Description: Office blood pressure measured at trough by automatic oscillometric device.
Time Frame: Change from Baseline Visit 1 (week 0) to Visit 4 (Week 6)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 288 | 139
mm Hg | -18.2 (16.7) | -12.3 (17.7)

2. Primary Outcome: Change From Baseline in Mean Seated Diastolic Blood Pressure After 6 Weeks of Nebivolol Monotherapy
Description: Office blood pressure measured at trough by automatic oscillometric device.
Time Frame: Change from Baseline (Week 0) to Visit 4 (Week 6)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 288 | 139
mm Hg | -12.3 (9.8) | -5.7 (11.4)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for a period of 10 months, from March 2010 to January 2011.
Arm/Group | Nebivolol | Placebo
Serious Adverse Events (participants affected / at risk) | 1/290 | 3/142
Other Adverse Events (participants affected / at risk) | 0/290 | 0/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol (N=290) | Placebo (N=142)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.